CLINICAL TRIAL: NCT01603914
Title: Comparison of Three Strategies for Changing of Central Venous Catheters in Patients With Serious Burns for the Prevention of Catheter-associated Bacteremia: Randomized Clinical Trial
Brief Title: Central Venous Catheter Replacement Strategies in Adult Patients With Major Burn Injury
Acronym: CARB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Oscar Penuelas, MD, MD, Attending of Critica Care Department and Burns Center, Hospital Universitario de Getafe, Hospital Universitario Getafe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI11/01121; ISCIII (Other Grant/Funding Number: Instituto de Salud Carlos III. Ministerio de Economía, Spain)
Record Dates: First submitted 2012-05-13; First posted 2012-05-23 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-05

CONDITIONS: Catheter-related Bloodstream Infection; Complication of Catheter
Keywords: burns, catheter related bacteremia,; infection, central venous catheter,; catheter-related bloodstream, adult critically ill patients
MeSH Terms: conditions — Burns; Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- scheduled wire-guided every six days (Experimental): scheduled wire-guided every six days and a replacement of the catheter in a different place after 12 days from randomization.
  Interventions: Device: central venous catheter replacement (Arrowgard Blue plus Quad-Lumen CVC )
- Scheduled replacement every six days (Experimental): Scheduled replacement every six days in a different location
  Interventions: Device: central venous catheter replacement (Arrowgard Blue plus Quad-Lumen CVC )
- replacement guided by clinical criteria (Experimental): re change of catheter strategy guided by clinical suspicious of catheter-related bacteremia and replacement of the catheter in a different location.
  Interventions: Device: central venous catheter replacement (Arrowgard Blue plus Quad-Lumen CVC )

INTERVENTIONS:
Device: central venous catheter replacement (Arrowgard Blue plus Quad-Lumen CVC ) — Routine practices for the type of catheter of each participating Unit will be respected. Multilumen central venous catheter will be used (i.e Arrowgard Blue plus Quad-Lumen CVC set). Impregnated Catheter with antiseptics or with antibiotics will be allowed.The anatomical locations selected for the replacement of central venous catheter are: subclavian vein, internal jugular vein, femoral vein and the change will be addressed according to the randomization.
  The dressing and maintenance of the catheter will be guided according with the Guides of The Centers for Disease Control and Prevention (CDCs) and a check-in lists will be fill in for each catheter.
  A pre-defined stratified analysis will be performed according with: type of catheter, participating unit, and insertion site.
  Other Names: Catheter Related Bacteremia in Burns, CARBB study

SUMMARY:
The aim of this project is to answer the following questions:

To determine the incidence of catheter related bacteremia (CRB) with three strategies of central venous catheter exchange in critically ill adult patients with major burn and to determine the regimen that will minimize the risk of bacteremia.

To determine the incidence rate of catheter colonization in adult patients with major burns.

The scientific knowledge to be acquired through this project is of likely benefit to the care of critically ill patients with burns injury as follows:

The intention is to improve the outcomes in critically ill patients by minimizing one of the most frequent causes of infection in the Burn Intensive Care Unit, those from central venous catheters. Decreasing infections will decrease morbidity, decrease length of stay, decrease costs, and decrease mortality.

DETAILED DESCRIPTION:
Aim: To determine the incidence of catheter-related bacteremia (CRB) with three primary schedules of central venous catheter exchange in adult critically ill patients with major burn injury.

Hypothesis: A strategy of catheter exchange according with clinical criteria will result in no more CRB compared with a routine catheter changes without guidewire exchange strategy or frequent guidewire exchange or frequent new-site replacement.

Background: The intravenous catheter-related bacteremia (ICRB) is a nosocomial infection affecting patients admitted to intensive care and that leads to increased morbidity. Accumulative incidence rates of ICRB are 5.5 infections per 1000 catheters-day. Several strategies have been proposed to decrease of the rate of ICRB in critically ill patients. However, there is not agreement to recommend a replacement pattern of central venous catheters in adult critically ill patients with major burns as a strategy for the reduction in intravenous catheter-associated bacteremia.

Objectives. To compare three strategies of replacement from central venous catheters for the prevention of ICRB. Find out the risk of mechanical complications associated with each strategy of central venous catheter replacement.

Method. Randomized, multicenter clinical trial, single blind to compare three strategies for intravenous catheter replacement in patients with major burns: a scheduled wire-guided strategy every six days: second, a scheduled strategy of replacement every six days in a different punction and third, a re-change strategy guided by clinical criteria for suspicion of catheter-associated infection. Primary outcome: catheter colonization rate and rate of intravenous catheter-associated bacteremia. Secondarily, we calculate the incidence rate of colonization of central venous catheter and finally we will analyze the associated complications.

This project requires enough patients to show a difference between three intervention groups. A significant decrease in infection rate would be from the current 20 infections per 1000 catheter days to approximately 15 per 1000 catheter days. This would require a minimum of 1000 catheter days per group.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old) admitted in a Critical Care Burn Center with a total body surface area (TBSA) greater than 20% and/or smoke inhalation injury.

Exclusion Criteria:

* Adults admitted in a Critical Care Burn Center with a Do-Not-Resuscitate (DNAR) order due to severity of injuries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Accumulative Incidence rate of catheter-related bacteremia | participants will be followed for the duration of Burn Center stay, an expected lenght of stay average of 6 weeks (that represents the mean length of stay average in our BUrn Center in 2011)

SECONDARY OUTCOMES:
Accumulative incidence rate of catheter colonization | participants will be followed for the duration of Burn Center stay, an expected lenght of stay average of 6 weeks (that represents the mean length of stay average in our BUrn Center in 2011)
  From date of randomization until the date of first documented progression or date of adverse event (pneumothorax, hemothorax)or death from any cause, whichever came first, assessed up to 18 months.
Mechanical complications of catheter insertion | during the procedure of central catheter insertion
  Neumothorax, hemothorax, arterial puncture,

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Penuelas, MD, Principal Investigator — Critical Care Department and Burn Center. Hospital Universitario de Getafe, Madrid, Spain
Locations (3):
- Spain (3):
  - Complejo Hospitalario Universitario de A Coruna, A Coruña, A Coruna
  - Critical Care and Burn Unit, Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital de Cruces, Barakaldo, Vizcaya

REFERENCES:
- [Background] Silver GM, Klein MB, Herndon DN, Gamelli RL, Gibran NS, Altstein L, McDonald-Smith GP, Tompkins RG, Hunt JL; Inflammation and the Host Response to Trauma, Collaborative Research Program. Standard operating procedures for the clinical management of patients enrolled in a prospective study of Inflammation and the Host Response to Thermal Injury. J Burn Care Res. 2007 Mar-Apr;28(2):222-30. doi: 10.1097/BCR.0B013E318031AA44. PMID 17351437
- [Result] O'Mara MS, Reed NL, Palmieri TL, Greenhalgh DG. Central venous catheter infections in burn patients with scheduled catheter exchange and replacement. J Surg Res. 2007 Oct;142(2):341-50. doi: 10.1016/j.jss.2007.03.063. Epub 2007 Jul 12. PMID 17631903
- [Result] Brun-Buisson C, Doyon F, Sollet JP, Cochard JF, Cohen Y, Nitenberg G. Prevention of intravascular catheter-related infection with newer chlorhexidine-silver sulfadiazine-coated catheters: a randomized controlled trial. Intensive Care Med. 2004 May;30(5):837-43. doi: 10.1007/s00134-004-2221-9. Epub 2004 Apr 2. PMID 15060765
- See also: The American Burn Association is dedicated to improving the lives of everyone affected by burn injury through patient care, education, research and advocacy. — http://www.ameriburn.org/